CLINICAL TRIAL: NCT02395848
Title: Prospective, Open-label Trial to Evaluate Efficacy of 30-day Duration of Fidaxomicin in Patients With Recurrent C. Difficile Infection
Brief Title: Efficacy of 30-day Duration of Fidaxomicin for Recurrent C. Difficile Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient resource to complete the study
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDI.FIDAXOMICIN.1
Record Dates: First submitted 2015-02-26; First posted 2015-03-24 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-06

CONDITIONS: Clostridium Difficile Infection
Keywords: recurrent; infection
MeSH Terms: conditions — Clostridium Infections; Recurrence; Infections | interventions — Fidaxomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fidaxomicin (Experimental): 30-day Fidaxomicin ( 200mg twice daily x 10 days and 200mg once daily x 20 days.
  Interventions: Drug: Fidaxomicin

INTERVENTIONS:
Drug: Fidaxomicin — 200mg twice daily for 10 days followed by 200mg once daily for 20 days to prevent future recurrence of CDI
  Other Names: Dificid

SUMMARY:
This is a medical research study designed to look at the safety and efficacy of 30-day course of fidaxomicin for treatment of recurrent CDI (Clostridium difficile Infection). CDI is an infection that results when the normal flora (resident bacteria) of the colon is substantially altered by antibiotic treatment. The decrease in this normal flora allows for the growth of the C. difficile bacteria. Fidaxomicin is an antibiotic which is approved by Health Canada for treatment of CDI. Only patients with a primary case of CDI or 1st episode of recurrent CDI have been studied using a 10-day course of fidaxomicin.

DETAILED DESCRIPTION:
Clostridium difficile (C. difficile) infection (CDI) is one of the most frequent causes of healthcare associated infections and its rates are also growing in the community. The efficacy of standard antibiotics especially for recurrent CDI is limited as oral vancomycin and metronidazole also suppress the growth of anaerobic bacteria such as Bacteroides fragilis group which protect against proliferation of C. difficile. In contrast, in vitro study has shown that fidaxomicin has negligible activity against B. fragilis. The persistent disruption of healthy colonic flora may be the reason for recurrences following a course of treatment with metronidazole or vancomycin. Fidaxomicin has shown to reduce recurrences by approximately 50% when compared to oral vancomycin for primary or 1st episode of recurrent CDI.

Determining the efficacy and safety of 30-day duration of fidaxomicin for recurrent CDI through an open label clinical trial has important implications for policy making related to the drug reimbursement programs. In addition, the results of this study will be instrumental in demonstrating to the scientific and healthcare communities there may be a role for the 30-day course of fidaxomicin as a treatment modality for recurrent CDI. Curing CDI will restore the health and quality of life not just at the individual patient level but to the healthcare communities as well. Patients with refractory CDI require prolonged hospital admission, which increases the organism burden within the healthcare facilities. This in turn leads to the spread of the infection to other vulnerable patients. If a 30-day course of fidaxomicin proves to be safe and effective in curing patients with recurrent CDI, it will reduce the risk of severe complications in each patient and reduce transmission of CDI to other susceptible patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Able to provide informed consent.
3. Willing and able to comply with all the required study procedures.
4. A positive stool test for C. difficile toxin/gene using either PCR or enzyme immunoassay within 3 months of recruitment.
5. History of at least ≥ 2 recurrent CDI within 6 months where recurrence is deﬁned as return of diarrhea consistent with CDI within 8 weeks following CDI symptom resolution for at least 24 hours after a minimum of 10-day course of standard antibiotic therapy and positive stool test for C. difficile toxin or toxin gene and/or ongoing symptoms consistent with CDI despite at least 5 days of treatment using oral vancomycin.
6. Has more than three unformed bowel movements or 200 mL of stool for individuals with a stool collection device such as rectal tube or colostomy during a 24-hour period at the time of initiation of fidaxomicin. Participants will be enrolled when they meet inclusion criteria 1 - 5; will be initiated at fidaxomicin when they have CDI symptoms and stool will be tested for C. difficile toxin/gene. Only those with positive stool for C. difficile toxin/gene with current episode of CDI will continue with the study
7. Females of child bearing potential must be willing to use acceptable birth control as per the Health Canada Guidance Document: Considerations for Inclusion of Women in Clinical Trials and Analysis of Sex Differences.

Exclusion Criteria:

1. Planned or actively taking an investigational product for another study.
2. Prior fidaxomicin use.
3. Hypersensitivity to fidaxomicin or to any ingredient in the formulation or component of the container.
4. Evidence of toxic megacolon or gastrointestinal perforation on abdominal x-ray or life expectancy of less than 72 hours.
5. Active gastroenteritis due to Salmonella, Shigella, shiga toxin-producing E. coli, Yersinia or Campylobacter.
6. Anticipated requirement for systemic antibiotic therapy for more than 7 days during the study period.
7. Actively taking Saccharomyces boulardii or other probiotics other than yogurt.
8. Any condition that, in the opinion of the investigator, that the treatment may pose a health risk to the subject.
9. Pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07; Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine H Lee, MD, Principal Investigator — Vancouver Island Health Authority
Locations (1):
- Christine Lee, Victoria, BC - British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Fidaxomicin: 30-day fidaxomicin (200mg twice daily x 10 days followed by 200mg once daily x 20 days)
Period: Overall Study
Arm/Group | Fidaxomicin
Started | 31
Completed | 29
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Fidaxomicin: 30-day fidaxomicin
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 31

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at 30-day Completion of Fidaxomicin
Description: clinical response will be defined as those participants who have improvement in the number of bowel movements as determined by ≤ 3 unformed stools in a 24-hour period for 2 consecutive days during treatment and remaining well through study day 30.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 29
Participants | 24

2. Primary Outcome: Sustained Clinical Response 8 Weeks Following Completion of 30-day Course of Fidaxomicin
Description: sustained clinical response will be defined as those participants who have improvement in the number of bowel movements as determined by ≤ 3 unformed stools in a 24-hour period for 2 consecutive days during treatment and remaining well 8 weeks following completion of fidaxomicin
Time Frame: 8 week following completion of fidaxomicin
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 29
Participants | 22

3. Primary Outcome: Treatment Failure
Description: patients not meeting the definition of cure and requiring additional antibiotics for current CDI episode
Time Frame: Up to 8 weeks following completion of fidaxomicin
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Failure Requiring Additional Treatment for Recurrent C Difficile Infection: Number of participants requiring additional treatment for recurrent C. difficile infection within 8 weeks following completion of fidaxomicin
Arm/Group | Treatment Failure Requiring Additional Treatment for Recurrent C Difficile Infection
Number analyzed (Participants) | 29
Participants | 7

ADVERSE EVENTS:
Time Frame: Up to 8 weeks from the last dose of fidaxomicin; 12 weeks from enrollment into the study
Arm/Group | Fidaxomicin
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 2/29
Other Adverse Events (participants affected / at risk) | 7/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=29)
Clostridium difficile infection (Gastrointestinal disorders) | 1 (1)
Electrolyte disorder and uremia in a patient with pre-existing renal failure on chronic hemodialysis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=29)
Diarrhea (Gastrointestinal disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT02395848/Prot_SAP_000.pdf